CLINICAL TRIAL: NCT06026436
Title: Evaluation of the Effectiveness of Platelet-based and Microvesicle-based Assays to Predict Thrombotic and Bleeding Risk in Chronic Kidney Disease Patients With Acute Coronary Syndrome
Acronym: INNOV CKD 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM23_0073 - INNOV-CKD1
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease stage3
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CKD patients (Experimental)
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — 12-24 hours after P2Y12 ADP receptor loading dose (LD)
Biological: Blood samples — 1 month after Percutaneous Coronary Intervention (PCI)

SUMMARY:
This study is part of the RHU INNOV-CKD, winner of the 2019 call for projects. Its aim is to develop two biomarker assays to assess the thrombotic and haemorrhagic risks in patients with stage 3A or more severe chronic kidney disease (CKD) treated with percutaneous coronary intervention (PCI) and antiplatelet therapy following an acute coronary syndrome (ACS). We believe that these tests will help to adapt antiplatelet therapy on an individual basis (in terms of intensity and duration of treatment) and thus reduce the risk of thrombotic and haemorrhagic events in this particularly fragile population. The first biomarker corresponds to an intra-platelet molecule, Rap1b in its active form (known as aRap1b). The second is the pro-antithrombotic balance of circulating endothelial microvesicles (patEMV), which reflects endothelial dysfunction. An automated method for measuring these biomarkers will be developed in partnership with the D.Stago and BioCytex industries during the course of the project.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥18 years old and <90
* If the subject is a woman, she must be on contraception or menopausal.
* Non-ST-segment elevation ACS defined by the presence of at least 2 of the following criteria: (1) symptoms of myocardial ischemia, (2) electrocardiographic ST-segment abnormalities (depression or transient elevation of at least 0.1 mV) or T-wave inversion in at least in 2 contiguous leads, or (3) an elevated cardiac troponin value (above the upper limit of normal) 56 or ST segment elevation ACS scheduled for primary PCI defined 57 as a history of chest discomfort or ischemic symptoms of >20 minutes duration at rest ≤14 days prior to entry into the study with one of the following present on at least one ECG:

  1. ST-segment elevation ≥1 mm in two or more contiguous ECG leads
  2. New or presumably new left bundle branch block (LBBB).
  3. ST-segment depression ≥1 mm in two anterior precordial leads (V1 through V4) with clinical history and evidence suggestive of true posterior infarction
* Subject intended for an invasive strategy if NSTE-ACS or primary PCI if STE-ACS according to guidelines (appendix X)
* Subject with CKD stage 3A or higher (estimated glomerular filtration rate (eGFR) ≤ 60 ml/min/1.73 m2 according to the CKD-EPI formula
* Because of the documented biological variability of eGRF levels, patients with a eGRF < 78 ml/min/1.73 m2 can be included in this study, based on previous blood test results and on the investigator's decision. The DFG level of 78 ml/min/1.73 m2 correspond to an increase of 30 % of a DFG of 60 ml/min/1.73 m2. Indeed, the literature estimated a DFG levels variability of 30 % 58-61.
* Must be enrolled at a cardiac catheterization laboratory hospital or at a hospital/ambulance service affiliated with a cardiac catheterization laboratory hospital.
* Subject affiliated to or beneficiary of a social security system.
* Subject having signed written informed consent.

Exclusion Criteria:

* - Minors, pregnant or breast-feeding women;
* Subject under chronic anticoagulant
* Subject with thrombolytic therapy during the preceding 24 hours;
* Subject with bleeding diathesis;
* Subject not agreeing to participate.
* Subject with contraindication to clopidogrel, ticagrelor or to another anti platelet agent.
* Severe hepatic failure
* Ischemic Stroke within one month or a history of hemorrhagic stroke
* Platelet count<100 000
* Major surgery or trauma within 10 days
* Life expectancy <1 year
* Known significant bleeding risk according to the physician judgment
* Adults subject to a legal protection measure or unable to express their consent (persons under guardianship, curatorship or safeguard of justice)
* Persons deprived of their rights of liberty by judicial or administrative decision (persons in a situation of social fragility)
* Progressive cancer
* Systemic autoimmune disease
* Chronic viral or bacterial infections
* Diabetes requiring insulin therapy
* Constitutional haemorrhagic syndrome
* Organ transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
assessing the predictive value of high aRap1b expression | 12 months
  after antiplatelet loading dose in the occurrence of MACE

SECONDARY OUTCOMES:
High Rap1b-GTP expression | 1 month
  after antiplatelet loading dose in the occurrence of MACE
High Rap1b-GTP expression | 6 months
  after antiplatelet loading dose in the occurrence of MACE
High Rap1b-GTP expression | 1 month
  after antiplatelet loading dose and after PCI in the occurrence of bleeding events
High Rap1b-GTP expression | 6 months
  after antiplatelet loading dose and after PCI in the occurrence of bleeding events
High Rap1b-GTP expression | 12 months
  after antiplatelet loading dose and after PCI in the occurrence of bleeding events
Low Rap1b-GTP expression | 1 month
  after antiplatelet loading dose and after PCI in the occurrence of MACE
Low Rap1b-GTP expression | 6 months
  after antiplatelet loading dose and after PCI in the occurrence of MACE
Low Rap1b-GTP expression | 12 months
  after antiplatelet loading dose and after PCI in the occurrence of MACE
Low Rap1b-GTP expression | 12 months
  after antiplatelet loading dose and after PCI in the occurrence of bleeding events
High MV procoagulant and profibrinolytic expressions | 1 month
  after antiplatelet loading dose and after PCI, in the occurrence of MACE
High MV procoagulant and profibrinolytic expressions | 6 months
  after antiplatelet loading dose and after PCI, in the occurrence of MACE
High MV procoagulant and profibrinolytic expressions | 12 months
  after antiplatelet loading dose and after PCI, in the occurrence of MACE
High MV procoagulant and profibrinolytic expressions | 6 months
  after antiplatelet loading dose and after PCI, in the occurrence of bleeding
High MV procoagulant and profibrinolytic expressions | 12 months
  after antiplatelet loading dose and after PCI, in the occurrence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIS CREMIEUX, Study Director — Assistance Publique Hopitaux Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France